CLINICAL TRIAL: NCT01570270
Title: Cheese Intake and Hypercholesterolemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliera Brotzu (Other)
Responsible Party: Principal Investigator, Stefano Pintus, Principal Investigator, Azienda Ospedaliera Brotzu
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CASU
Record Dates: First submitted 2012-03-23; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Endocannabinoids
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- regular cheese (Experimental): This study was a 3-week, randomized, single blind, controlled, cross over clinical trial. The subjects were randomly assigned to eat 90g/d of the control or enriched cheese for 3 weeks, with a cross over after 3 weeks of washout. The study included 5 visits: 2 screening/baseline visits at weeks -1 and 0, 1 end of intake of 90 g/d of cheese visit at week 3, 1 end of the first wash out visit at week 6, and 1 end of treatment after crossing over visit at week 9. T
  Interventions: Dietary Supplement: CLA enriched cheese

INTERVENTIONS:
Dietary Supplement: CLA enriched cheese — This study was a 3-week, randomized, single blind, controlled, cross over clinical trial, conducted at the State Hospital Brotzu in Cagliari, Italy. The subjects were randomly assigned to eat 90g/d of the control or enriched cheese for 3 weeks, with a cross over after 3 weeks of washout. The study included 5 visits: 2 screening/baseline visits at weeks -1 and 0, 1 end of intake of 90 g/d of cheese visit at week 3, 1 end of the first wash out visit at week 6, and 1 end of treatment after crossing over visit at week 9.

SUMMARY:
In this study the investigators aimed at verifying whether consumption of a sheep cheese, naturally enriched in alpha-lipoic acid (ALA), conjugated linoleic acid (CLA) and vaccenic acid (VA), would modify the plasma lipid and endocannabinoid profiles in mild hypercholesterolemic subjects.

ELIGIBILITY:
Inclusion Criteria:

* 42 adult volunteers (19 male and 23 female) with diagnosed mild hypercholesterolemia (total cholesterol 220-290 mg/dL),
* 30-60 years of age

Exclusion Criteria:

* Pregnant (or those planning to become pregnant during the study period) and lactating women were excluded;
* also individuals with a self-reported history of diabetes, inflammatory bowel disease, pancreatitis, gallbladder or biliary disease in the past 12 months, and lactose intolerance before the screening visit.
* In addition, those with a history of cancer (except non-melanoma skin cancer) in the 2 years before screening, or of any major trauma or surgical event within 3 months before screening, were not enrolled.
* Volunteers with the following characteristics were also excluded:

  * total cholesterol ≥ 300 mg/dL,
  * serum triglycerides ≥ 250 mg/dL or ≤ 200 mg/dL,
  * HDL ≥ 70mg/dL,
  * BMI ≥ 30, or
  * uncontrolled hypertension (systolic blood pressure ≥ 160 mm Hg or
  * diastolic blood pressure ≥ 100 mm Hg) at screening.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
modification of LDL-cholesterol levels | baseline and 3 weeks